CLINICAL TRIAL: NCT00918060
Title: Clinical Effects of Locally-delivered Gel Containing Camella Sinensis Extracts
Brief Title: Clinical Effects of Locally-delivered Gel Containing Camella Sinensis Extracts as an Adjunct in Peridontitis Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Kanyawat Rattanasuwan, Department of Oral Medicine, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA. No. MU-IRB 2008/153.0511
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gel a (Experimental)
  Interventions: Drug: Camella sinensis gel
- gel b (Placebo Comparator)
  Interventions: Drug: Camella sinensis gel

INTERVENTIONS:
Drug: Camella sinensis gel — clinical effect of locally-delivered gel between Camella sinensis and placebo

SUMMARY:
The purpose of this study is to evaluate clinical result including plaque index, gingival inflammation, bleeding score, pocket depth reduction and clinical attachment level gain after used locally-delivered gel containing Camella sinensis extracts as an adjunctive treatment in periodontal therapy

ELIGIBILITY:
Inclusion Criteria:

* subjects have sound tooth with pocket depth = or > 5 mm. without caries, restoration, mobility and furcation involvement
* no systemic complicated factors
* no allergy to green tea or product of green tea
* signing in informed consent form

Exclusion Criteria:

* smoking
* pregnancy or lactation
* antibiotic premedication or antibiotic intake in previous 3 month

Ages: 34 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
pocket depth reduction, clinical attachment level gain, gingival index, bleeding score | baseline, 1, 3 and 6 month after gel had loaded

SECONDARY OUTCOMES:
plaque index | baseline, 1, 3, and 6 month after gel had loaded

CONTACTS AND LOCATIONS:
Overall Officials: Kanyawat Rattanasuwan, Study Director — Department of Oral Medicine, Mahidol University; Kanyawat Rattanasuwan, Study Chair — Maha Chakri Sirindhorn Dental Hospital

REFERENCES:
- [Derived] Rattanasuwan K, Rassameemasmaung S, Sangalungkarn V, Komoltri C. Clinical effect of locally delivered gel containing green tea extract as an adjunct to non-surgical periodontal treatment. Odontology. 2016 Jan;104(1):89-97. doi: 10.1007/s10266-014-0190-1. Epub 2014 Dec 19. PMID 25523604